CLINICAL TRIAL: NCT07024992
Title: A National Test of a Culturally Tailored Smartphone-based Smoking Cessation and Mental Health Intervention for Black Adults With HIV
Brief Title: Enhancing Smoking Cessation for African American People Everywhere
Acronym: ESCAPE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Lorra Garey, Research Associate Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004985
Record Dates: First submitted 2025-05-05; First posted 2025-06-17 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: ESCAPE Intervention+NRT; quitSTART Intervention+NRT; CTRL+NRT
Keywords: HIV; Anxiety Sensitivity; Mobile Health; Smoking; Smoking Cessation; African American; Ecological Momentary Assessments; Just-in-Time Adaptive Intervention
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESCAPE intervention + NRT (Experimental)
  Interventions: Behavioral: ESCAPE app + NRT
- quitSTART intervention + NRT (Active Comparator)
  Interventions: Behavioral: quiSTART app + NRT
- Control (CTRL) (Sham Comparator)
  Interventions: Behavioral: Control (CTRL)

INTERVENTIONS:
Behavioral: ESCAPE app + NRT — ESCAPE is a mobile intervention that targets anxiety sensitivity among Black adults who smoke cigarettes and have HIV. This intervention is framed within the cultural context of interoceptive stress among Black adults who smoke, which is supported by theory, empirical evidence, and characteristics of this group. The intervention employs a variety of features to educate users on how to deal with stress, anxiety, and nicotine withdrawal symptoms. The app contains a series of on-demand features, including a coping toolkit, stress management trainings, and a series of educational videos. ESCAPE also utilizes Ecological Momentary Assessments (EMAs) to gather information and provide personalized messages to users in real time. All participants will receive free nicotine replacement therapy (NRT).
  Arms: ESCAPE intervention + NRT
Behavioral: quiSTART app + NRT — quitSTART is a smartphone-based National Cancer Institute (NCI) intervention for standard mobile smoking cessation treatment. The intervention contains features that allow its' users to better understand their smoking patterns, and build skills needed to become and stay smoke free. The app allows users to track cravings and delivers motivational messages to users for each craving they track. All participants will receive free nicotine replacement therapy (NRT).
  Arms: quitSTART intervention + NRT
Behavioral: Control (CTRL) — The CTRL group will complete the same baseline survey, follow-up surveys, and ecological momentary assessments as the ESCAPE app + NRT and the quitSTART app + NRT group. All participants will receive free nicotine replacement therapy (NRT). They will not receive additional intervention content.
  Arms: Control (CTRL)

SUMMARY:
The present study aims to investigate the efficacy of an mHealth smoking cessation and HIV disease management intervention among a nationally representative sample of African America/Black (hereafter refer to as Black) persons with HIV/AIDS (PWH) who smoke cigarettes. Participants will be randomized into one of three conditions: (1) the intervention, ESCAPE (Enhancing Smoking Cessation for African American People Everywhere) + Nicotine Replacement Medications (NRT), (2) the National Cancer Institute's (NCI) quitSTART app, the standard mobile smoking cessation treatment + NRT, and (3) an assessment-only control group + NRT.

DETAILED DESCRIPTION:
This nationwide trial aims to evaluate the efficacy of a smartphone-based smoking cessation and HIV care management intervention culturally tailored for Black PWH who smoke cigarettes with treated and untreated HIV.A RCT will be conducted with 300 Black PWH who smoke cigarettes to evaluate the efficacy of the intervention. Participants will be randomly assigned to the smartphone-based ESCAPE intervention + NRT, the National Cancer Institute's smartphone-based quitSTART intervention + NRT, or assessment-only control + NRT. Participants will complete a self-screener, baseline appointment, 8 weeks of ecological momentary assessments (2x per day; EMAs), 8 weekly follow-up assessments, 10 monthly check-in surveys, a 28-week follow-up, and a final 54-week follow-up. A subset of participants will also be selected to complete a qualitative interview at the end of their 6th week in the study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Identify as Black/African American
* Living with HIV
* Willing and able to complete study assessments
* Smoking at least 5 cigarettes per day for at least a year
* Motivated to quit smoking (≥ 5 on a 10-point scale)
* Must be ready to quit cigarettes within 14 days of full enrollment
* Moderate or higher anxiety sensitivity (i.e., ≥ 5 on the Short Scale Anxiety Sensitivity Index [SSASI]) OR elevated anxiety (i.e., > 7 on the Overall Anxiety Severity and Impairment Scale [OASIS]) OR depression (i.e., > 7 on the Overall Depression Severity and Impairment Scale [ODSIS])
* Must be interested in using a mobile app
* Must be willing to download a mobile app onto their personal phone
* Must be willing to use NRT
* Possess an Android/Apple smartphone that is compatible with the mobile app
* Demonstrate 7th grade level proficiency in English (> 4 on the Rapid Estimate of Adult Literacy in Medicine-Short Form [REALM-SF])
* Valid proof of identification (photo of valid US ID)

Exclusion Criteria:

* Legal situations which may interfere with study participation
* Not being fluent in English
* High blood pressure that is not under control
* Having experienced a heart attack within the past 2 weeks
* Pregnant of planning to become pregnant within the next six months
* Cognitive impairment (a score of > 8 on the Six-Item Cognitive Impairment Test [6-CIT])
* Residing in a location (Urban/Rural) for which the corresponding study cell has been filled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-05-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
7-day Biochemically Verified Point Prevalence Abstinence (PPA) | Collected during the 54-week follow-up assessment
  PPA will be defined as no cigarette smoking within the past 7 days, and will be biochemically verified via assessment of expired carbon monoxide (< 6 ppm).
Anxiety | Baseline appointment through the 54-week follow-up, inclusive of follow-up assessments (Weeks 1-6, 28, and 54-week)
  Anxiety will be evaluated via Overall Anxiety Severity Index Scale (OASIS).
Depression | Baseline appointment through the 54-week follow-up, inclusive of follow-up assessments (Weeks 1-6, 28, and 54-week).
  Depression will be evaluated via the Overall Depression Severity Index Scale (ODSIS).
HIV (and general) Quality of Life | Baseline appointment through the 54-week follow-up, inclusive of every assessment containing these survey items (daily 3x EMAs for 8 weeks and weeks 1-6, 28, and 54-week follow-ups)
  HIV (and general) quality of life will be evaluated using continuous variables (e.g., the World Health Organization HIV Quality of Life Brief Scale, the Quality of Life Enjoyment and Satisfaction Questionnaire, and the Index of Engagement in HIV Care).
HIV Care Adherence/Engagement | Baseline appointment through the 54-week follow-up, inclusive of every assessment containing these survey items (daily 3x EMAs for 8 weeks and weeks 1-6, 28, and 54-week follow-ups)
  HIV-related outcomes will be evaluated using the dichotomous variables (e.g., ART medication non-adherence and missed treatment appointments).

SECONDARY OUTCOMES:
Anxiety Sensitivity Reduction | Baseline appointment through the 54-week follow-up, inclusive of follow-up assessments (Weeks 1-6, 28, and 54-week)
  Anxiety sensitivity will be evaluated using the Short Scale Anxiety Sensitivity Index (SSASI).

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Businelle, Ph.D., Principal Investigator — University of Oklahoma Health Sciences
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be uploaded to the National Institutes of Health National Data Archive where it can be accessed by other researchers who have uploaded to the National Data Archive.
Time Frame: 1 year from completion of aims of the project (i.e., publication of the main outcome paper)
Access Criteria: The data can be accessed by researchers who request access to the data and complete a Data use Certification (DUC), certifying that have a research need related to the data.